CLINICAL TRIAL: NCT03845257
Title: Correlation of FeNO, Blood Eosinophils, Bronchoalveolar Lavage Findings and Bronchial Epithelium Histopathology in Patients With Chronic Obstructive Pulmonary Disease and Asthma
Status: Terminated | Type: Observational
Why Stopped: difficult patient recruitment
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Daniela Gompelmann, Daniela Gompelmann, MD, Heidelberg University
Other Study IDs: Protocol DG3.0 - 25.06.2018
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Lung Diseases
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Blood Specimen Collection; Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COPD: The following parameters are to be evaluated:
  * Blood eosinophils
  * FeNO
  * Eosinophils in bronchoalveolar lavage
  * Tissue eosinophilia (protected specimen brush sampling, endobronchial biopsy)
  Interventions: Diagnostic Test: Blood sampling, FeNO, bronchoalveolar lavage, bronchoscopic tissue sampling
- Patients with asthma: The following parameters are to be evaluated:
  * Blood eosinophils
  * FeNO
  * Eosinophils in bronchoalveolar lavage
  * Tissue eosinophilia (protected specimen brush sampling, endobronchial biopsy)
  Interventions: Diagnostic Test: Blood sampling, FeNO, bronchoalveolar lavage, bronchoscopic tissue sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling, FeNO, bronchoalveolar lavage, bronchoscopic tissue sampling — Blood sampling (eosinophil count; eosinophilia is defined as >300/µl (or >150/µl during oral glucocorticosteroid treatment); FeNO: Measurement of fractional nitric oxide (NO) concentration in exhaled breath; Bronchoscopy: BAL: total leukocyte counts and leukocyte differential counts including eosinophils, PSB sampling: eosinophil count/100 cells, endobrochial biopsy: tissue eosinophil count/100 cells.

SUMMARY:
Scientific research focuses on "eosinophilic inflammation" as it seems to guide the therapeutic regimen in patients with asthma and COPD. The primary objective of this prospective trial is to evaluate which parameter(s) best reflects eosinophilic inflammation by correlating tissue eosinophils (endobronchial biopsy, protected specimen brush sampling) with FeNO, peripheral blood eosinophils, and eosinophils in the bronchoalveolar lavage of patients with obstructive pulmonary disease.

DETAILED DESCRIPTION:
This is a multicenter prospective trial. Enrollment will continue until 150 patients with chronic obstructive pulmonary disease and 50 patients with severe asthma have been entered into this trial and have completed bronchoscopic evaluation. In this trial, the following parameters are to be evaluated:

* Blood eosinophils (absolute and relative)
* FeNO
* Eosinophils in bronchoalveolar lavage
* Tissue eosinophilia (protected specimen brush sampling, endobronchial biopsy)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of COPD or asthma (according to the guidelines)
* Age >18 years
* Indication for bronchoscopy for medical reasons (not study-related)
* Ability to provide informed consent

Exclusion Criteria:

* paO2 <60 mmHg on 4L 02 /min, paCO2 > 55 mmHg on room air
* FEV1 <20%
* Pulmonary infection or exacerbation within the last 4 weeks
* Additional pulmonary diseases (pneumonia, lung cancer, tuberculosis, interstitial lung disease)
* Contraindication for BAL, PSB sampling or endobronchial biopsy
* Current use of anticoagulants that can not be stopped for bronchoscopy
* Heart failure with left ventricular ejection fraction <30%
* Myocardial infarction in previous 6 months
* Significant pulmonary hypertension (PAPS >45 mmHg, right heart failure [echocardiography] and/or PAPm >35 mmHg [right heart catheter])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of COPD or asthma (according to the guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Assessment of eosinophilic inflammation by correlating tissue eosinophilia with eosinophil count in blood/BAL and FeNO measurement. | 18 months
  Correlation of FeNO, blood eosinophils, bronchoalveolar lavage findings and bronchial epithelium histopathology in patients with chronic obstructive pulmonary disease and asthma

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gompelmann, Principal Investigator — Thoraxklinik University Heidelberg
Locations (3):
- Macquarie University Sydney, Sydney, New South Wales, Australia
- Germany (2):
  - Division of Clinical Infectious Diseases/Research Center Borstel, Borstel
  - Thoraxklinik University Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: Undecided